CLINICAL TRIAL: NCT04317872
Title: Do Peri-operative High Doses of Intravenous Glucocorticoids Improve Short-term Functional Outcome After Direct Anterior Total Hip Arthroplasty? A Randomized, Single Surgeon, Placebo Controlled, Double Blind Study
Brief Title: Effect of Peri-operative Glucocorticoids on Short-term Functional Outcome After THA
Acronym: DEXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S63584
Record Dates: First submitted 2020-03-17; First posted 2020-03-23 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Coxarthrosis; Avascular Necrosis of Hip
Keywords: Total Hip Arthroplasty; Direct Anterior Approach; Glucocorticoids; Short term functional outcome
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: A randomized, single surgeon, placebo controlled, double blind study using two parallel study groups
Who Masked: Participant, Care Provider
Masking Description: An anesthetist or study nurse not involved in further care of the patient nor in the study will prepare the medication to administered based on the allocated group. The first syringe with either 5 or 25 mg of Aacidexam will be administered during induction. The second syringe will go with the patient to the ward and will be administered 12 hours after the surgery by the (blinded) ward nurse. The patient will not be made aware of what has been administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Current protocol (Experimental): "Current protocol": patients will receive a single shot of 25mg of aacidexam iv (5cc) at induction. After 12 hours these patients will another shot of 10mg of aacidexam iv (2cc) on the ward.
  Interventions: Drug: High dose of peri-operative intravenous dexamethasone
- Old protocol (Active Comparator): "Old protocol": patients will receive a single shot of 5mg of aacidexam iv at induction (5cc). After arrival 12 hours these patients will receive a placebo, i.e. a shot of 2 cc of NaCl 0.9% iv (Mini-Plasco van B. Braun).
  Interventions: Drug: Low dose of peri-operative intravenous dexamethasone

INTERVENTIONS:
Drug: High dose of peri-operative intravenous dexamethasone — 25mg aacidexam is administered during induction followed by 10mg on the ward after 12 hours
  Other Names: Aacidexam
  Arms: Current protocol
Drug: Low dose of peri-operative intravenous dexamethasone — 10mg aacidexam is administered during induction followed by placebo on the ward after 12 hours
  Other Names: Aacidexam
  Arms: Old protocol

SUMMARY:
This randomized, single surgeon, placebo controlled, double blind study will be conducted in order to investigate whether or not peri-operative high doses of intravenous glucocorticoids improve short-term functional outcome after direct anterior total hip arthroplasty. So far, it has been proven that high dose glucocorticoids reduce immediate post-operative pain and nausea, but no data exists on functional outcome during the first 6 weeks. Our hypothesis is that patients in the intervention group will follow a so-called "get ahead, stay ahead" principle and that glucocorticoids can be considered an important tool (adjuvant treatment) in the enhanced recovery pathway after THA with significant socio-economic implications.

DETAILED DESCRIPTION:
Patients listed for a direct anterior total hip arthroplasty by a single surgeon will be recruited for this study and allocated to one of two groups:

1. intervention group: 25 grams of iv dexamethasone at induction followed by 10 mg of iv dexamethasone 12 hours later
2. control group: 5 grams of iv dexamethasone at induction followed by placebo 12 hours later Both patients and surgeons will be blinded. Primary outcome measure will be number of steps during the first 6 weeks as measured by a pedometer. Secondary outcome measures will be side effects, complications, Patient Reported Outcome Measures, pain, nausea, stiffness, achievement of clinical milestones and use of analgesia/anti-emetics. This data will be collected using a tailor made application for a smartphone or tablet and data collecting will start one week before surgery until 6 weeks after surgery.

Based on a power analysis both groups will consist of 35 patients each.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing unilateral uncemented THA for primary OA or AVN of the hip under general anesthesia (GA)
* Aged 18 years and above (including women of child bearing age)
* Able to provide informed consent

Exclusion Criteria:

* Younger than 18 years
* Known alcohol or drug abuse
* Known allergy for glucocorticoids
* Administration of any glucocorticoids in the last three months
* Usage of strong analgesia (such as lyrica or oxycodone) as regular medication
* Usage of medication with anticipated interactions with glucocorticoids
* Known gastric ulcer
* Insulin dependent diabetes mellitus
* Severe heart disease (NYHA > 2)
* Liver or renal failure
* Systemic rheumatoid diseases
* Insufficient understanding of the Dutch language
* Unable to provide informed consent
* Pre-operative use of walking aids
* Gross anatomical deformities
* Significant intra-operative complications such as periprosthetic fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Steps | 6 weeks
  Number of steps as measured by a pedometer

SECONDARY OUTCOMES:
Post-operative nausea and vomiting | up to 1 week, 0-10, lower scores indicate better clinical outcome
  Post-operative nausea and vomiting Visual Analogue Scale scores
Same day mobilization | 1 day (yes or no)
  Whether or not if was possible for the physiotherapists to mobilize the patient on the day of surgery
Clinical milestones | 6 weeks
  Time to achieve certain clinical milestones, e.g. climbing stairs, driving a car, etc
Oxford Hip Score | 6 weeks
  Patients Reported Outcome Measures
Western Ontario and McMaster Universities Osteoarthritis Index | 6 weeks
  Patients Reported Outcome Measures
Hip dysfunction and Osteoarthritis Outcome Score | 6 weeks
  Patients Reported Outcome Measures
Forgotten Joint Score | 6 weeks
  Patients Reported Outcome Measures
Short Form 36 | 6 weeks
  Patients Reported Outcome Measures
Fatigue Severity Scale | 6 weeks
  Patients Reported Outcome Measures
Groningen Activity Restriction Scale | 6 weeks
  Patients Reported Outcome Measures
Pain scores | 6 weeks, 0-10, lower scores indicate better clinical outcome
  Visual Analogue Scale scores during the day, the night and during exercises
Stiffness | 6 weeks, 0-10, lower scores indicate better clinical outcome
  Visual Analogue Scale scores
Use of Analgesia | 6 weeks
  The use of analgesia such as paracetamol (acetominophen), NSAIDs, and morphine(like) substances
Use of Anti-emetics | Up to 1 week
  The use anti-emetics to reduce direct post-operative nausea
Complications | 6 weeks
  The occurrence of complications such as wound healing problems, infections, allergic reactions, venous thrombo-embolisms, etc
Side effects | 6 weeks
  The occurrence of side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Ghijselings, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Marques EM, Jones HE, Elvers KT, Pyke M, Blom AW, Beswick AD. Local anaesthetic infiltration for peri-operative pain control in total hip and knee replacement: systematic review and meta-analyses of short- and long-term effectiveness. BMC Musculoskelet Disord. 2014 Jul 5;15:220. doi: 10.1186/1471-2474-15-220. PMID 24996539
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] Choi PT, Bhandari M, Scott J, Douketis J. Epidural analgesia for pain relief following hip or knee replacement. Cochrane Database Syst Rev. 2003;2003(3):CD003071. doi: 10.1002/14651858.CD003071. PMID 12917945
- [Background] Moskal JT, Capps SG. Meta-analysis of Intravenous Tranexamic Acid in Primary Total Hip Arthroplasty. Orthopedics. 2016 Sep 1;39(5):e883-92. doi: 10.3928/01477447-20160526-02. Epub 2016 Jun 1. PMID 27248332
- [Background] Hojer Karlsen AP, Geisler A, Petersen PL, Mathiesen O, Dahl JB. Postoperative pain treatment after total hip arthroplasty: a systematic review. Pain. 2015 Jan;156(1):8-30. doi: 10.1016/j.pain.0000000000000003. PMID 25599296
- [Background] Nanni M, Perna F, Calamelli C, Donati D, Ferrara O, Parlato A, D'Arienzo M, Faldini C. Wound drainages in total hip arthroplasty: to use or not to use? Review of the literature on current practice. Musculoskelet Surg. 2013 Aug;97(2):101-7. doi: 10.1007/s12306-013-0270-3. Epub 2013 May 25. PMID 23709186
- [Background] Villatte G, Mathonnet M, Villeminot J, Savary M, Theissen A, Ostermann S, Erivan R, Raynaud-Simon A, Slim K. [Interest of enhanced recovery programs in the elderly during total hip arthroplasty A systematic review]. Geriatr Psychol Neuropsychiatr Vieil. 2019 Sep 1;17(3):234-242. doi: 10.1684/pnv.2019.0796. French. PMID 31251213
- [Background] Kardash KJ, Sarrazin F, Tessler MJ, Velly AM. Single-dose dexamethasone reduces dynamic pain after total hip arthroplasty. Anesth Analg. 2008 Apr;106(4):1253-7, table of contents. doi: 10.1213/ANE.0b013e318164f319. PMID 18349202
- [Background] Mathiesen O, Jacobsen LS, Holm HE, Randall S, Adamiec-Malmstroem L, Graungaard BK, Holst PE, Hilsted KL, Dahl JB. Pregabalin and dexamethasone for postoperative pain control: a randomized controlled study in hip arthroplasty. Br J Anaesth. 2008 Oct;101(4):535-41. doi: 10.1093/bja/aen215. Epub 2008 Jul 23. PMID 18653493
- [Background] Bergeron SG, Kardash KJ, Huk OL, Zukor DJ, Antoniou J. Perioperative dexamethasone does not affect functional outcome in total hip arthroplasty. Clin Orthop Relat Res. 2009 Jun;467(6):1463-7. doi: 10.1007/s11999-009-0733-x. Epub 2009 Feb 18. PMID 19224304
- [Background] Rasmussen ML, Mathiesen O, Dierking G, Christensen BV, Hilsted KL, Larsen TK, Dahl JB. Multimodal analgesia with gabapentin, ketamine and dexamethasone in combination with paracetamol and ketorolac after hip arthroplasty: a preliminary study. Eur J Anaesthesiol. 2010 Apr;27(4):324-30. doi: 10.1097/EJA.0b013e328331c71d. PMID 19734790
- [Background] Miyagawa Y, Ejiri M, Kuzuya T, Osada T, Ishiguro N, Yamada K. Methylprednisolone reduces postoperative nausea in total knee and hip arthroplasty. J Clin Pharm Ther. 2010 Dec;35(6):679-84. doi: 10.1111/j.1365-2710.2009.01141.x. PMID 21054459
- [Background] Jiang J, Wang H, Wang Y. [Clinical study on effect of dexamethasone in preventing fat embolism syndrome after cemented hip arthroplasty]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2010 Aug;24(8):913-6. Chinese. PMID 20839434
- [Background] Lunn TH, Kristensen BB, Andersen LO, Husted H, Otte KS, Gaarn-Larsen L, Kehlet H. Effect of high-dose preoperative methylprednisolone on pain and recovery after total knee arthroplasty: a randomized, placebo-controlled trial. Br J Anaesth. 2011 Feb;106(2):230-8. doi: 10.1093/bja/aeq333. Epub 2010 Dec 3. PMID 21131371
- [Background] Lunn TH, Andersen LO, Kristensen BB, Husted H, Gaarn-Larsen L, Bandholm T, Ladelund S, Kehlet H. Effect of high-dose preoperative methylprednisolone on recovery after total hip arthroplasty: a randomized, double-blind, placebo-controlled trial. Br J Anaesth. 2013 Jan;110(1):66-73. doi: 10.1093/bja/aes345. Epub 2012 Sep 17. PMID 22986420
- [Background] Backes JR, Bentley JC, Politi JR, Chambers BT. Dexamethasone reduces length of hospitalization and improves postoperative pain and nausea after total joint arthroplasty: a prospective, randomized controlled trial. J Arthroplasty. 2013 Sep;28(8 Suppl):11-7. doi: 10.1016/j.arth.2013.05.041. Epub 2013 Aug 9. PMID 23937923
- [Background] Koh IJ, Chang CB, Lee JH, Jeon YT, Kim TK. Preemptive low-dose dexamethasone reduces postoperative emesis and pain after TKA: a randomized controlled study. Clin Orthop Relat Res. 2013 Sep;471(9):3010-20. doi: 10.1007/s11999-013-3032-5. Epub 2013 May 4. PMID 23645340
- [Background] McLawhorn AS, Beathe J, YaDeau J, Buschiazzo V, Purdue PE, Ma Y, Sculco TP, Jules-Elysee K. Effects of steroids on thrombogenic markers in patients undergoing unilateral total knee arthroplasty: a prospective, double-blind, randomized controlled trial. J Orthop Res. 2015 Mar;33(3):412-6. doi: 10.1002/jor.22776. Epub 2015 Jan 6. PMID 25565656
- [Background] Sculco PK, Pagnano MW. Perioperative solutions for rapid recovery joint arthroplasty: get ahead and stay ahead. J Arthroplasty. 2015 Apr;30(4):518-20. doi: 10.1016/j.arth.2015.01.036. Epub 2015 Jan 30. PMID 25680452
- [Background] Xu B, Ma J, Huang Q, Huang ZY, Zhang SY, Pei FX. Erratum to: Two doses of low-dose perioperative dexamethasone improve the clinical outcome after total knee arthroplasty: a randomized controlled study. Knee Surg Sports Traumatol Arthrosc. 2018 Jun;26(6):1879. doi: 10.1007/s00167-017-4593-8. No abstract available. PMID 28631144
- [Background] Lei YT, Xu B, Xie XW, Xie JW, Huang Q, Pei FX. The efficacy and safety of two low-dose peri-operative dexamethasone on pain and recovery following total hip arthroplasty: a randomized controlled trial. Int Orthop. 2018 Mar;42(3):499-505. doi: 10.1007/s00264-017-3537-8. Epub 2017 Jun 25. PMID 28647788
- [Background] Lei Y, Huang Q, Xu B, Zhang S, Cao G, Pei F. Multiple Low-Dose Dexamethasone Further Improves Clinical Outcomes Following Total Hip Arthroplasty. J Arthroplasty. 2018 May;33(5):1426-1431. doi: 10.1016/j.arth.2017.11.057. Epub 2017 Dec 5. PMID 29258763
- [Background] Dissanayake R, Du HN, Robertson IK, Ogden K, Wiltshire K, Mulford JS. Does Dexamethasone Reduce Hospital Readiness for Discharge, Pain, Nausea, and Early Patient Satisfaction in Hip and Knee Arthroplasty? A Randomized, Controlled Trial. J Arthroplasty. 2018 Nov;33(11):3429-3436. doi: 10.1016/j.arth.2018.07.013. Epub 2018 Jul 19. PMID 30078660
- [Background] Toogood PA, Abdel MP, Spear JA, Cook SM, Cook DJ, Taunton MJ. The monitoring of activity at home after total hip arthroplasty. Bone Joint J. 2016 Nov;98-B(11):1450-1454. doi: 10.1302/0301-620X.98B11.BJJ-2016-0194.R1. PMID 27803219